CLINICAL TRIAL: NCT02536235
Title: Applied Topical Heat as an Adjunct for Pain Control in First-Trimester Surgical Abortion: A Randomized Controlled Trial
Brief Title: Applied Topical Heat as an Adjunct for Pain Control in First-Trimester Surgical Abortionl
Acronym: HAPPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Planned Parenthood of Greater New York (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SFPRF15-20
Record Dates: First submitted 2015-08-25; First posted 2015-08-31 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Topical Heat Application for Intraoperative Abortion Pain Management
MeSH Terms: interventions — Hot Temperature

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention: intraoperative topical heat (Experimental)
  Interventions: Other: heat
- Control: no intraoperative heat (No Intervention)

INTERVENTIONS:
Other: heat — activated heating pad to lower abdomen
  Arms: Intervention: intraoperative topical heat

SUMMARY:
Paracervical blocks are routinely used in first trimester surgical abortions and are a proven method for decreasing procedural pain. Even when paracervical anesthesia is used, an overwhelming majority of women still report at least moderate pain during a first trimester abortion procedure. Other than some non-pharmacologic modalities (music and visualization), only the addition of intravenous medication has been shown to reduce procedural pain. Applied topical heat is effective in alleviating pain in other medical subspecialties, and in gynecology has been shown to reduce pain from dysmenorrhea, but has never been studied for intraoperative pain control during first trimester abortion.

The investigators plan to conduct a double-blinded, randomized, controlled trial investigating the utility of topical heat application as an adjunct to paracervical block in first trimester surgical abortions up to 12 6/7wks. The primary outcome is pain score, measured using VAS, at time of uterine aspiration. As secondary outcomes, the investigators will look at the effect of heat application on pain at time of speculum placement, paracervical block, tenaculum placement, cervical dilation and overall pain. Patient satisfaction will also be assessed. If found to reduce pain during abortion under local anesthesia, the use of heat could offer an inexpensive, safe and universally available adjunct to the paracervical block during this procedure.

ELIGIBILITY:
Inclusion criteria

* Gestational age of 12 6/7 wks or less by ultrasound
* Age 16 years or older
* Requesting pregnancy termination by surgical abortion
* Eligible for outpatient pregnancy termination
* Able to provide informed consent
* English or Spanish* speaking *If research assistant hired for project is bilingual
* Electing local anesthesia only

Exclusion Criteria

* Reports active bleeding or severe pain at time of enrollment
* Early pregnancy failure identified on pre-operative ultrasound
* Skin irritation or rash over lower abdomen
* Presumed molar pregnancy
* Possible ectopic pregnancy
* Electing intravenous sedation
* Planned intra-operative sonographic guidance

Ages: 16 Years to 51 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2015-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
pain score measured on Visual Analog Scale (VAS) at time of uterine aspiration | collected at time of procedure.
  Level of pain at this step in the procedure will be recorded by patient on 100mm line where the left anchor point represents the absence of pain and the right anchor point represents the worst pain imaginable. The distance from the left anchor point to the patient's mark will be measured and recorded.

SECONDARY OUTCOMES:
pain score measured on VAS at time of speculum placement | collected at time of procedure.
  Level of pain at this step in the procedure will be recorded by patient on 100mm line where the left anchor point represents the absence of pain and the right anchor point represents the worst pain imaginable. The distance from the left anchor point to the patient's mark will be measured and recorded.
pain score measured on VAS at time of paracervical block | collected at time of procedure.
  Level of pain at this step in the procedure will be recorded by patient on 100mm line where the left anchor point represents the absence of pain and the right anchor point represents the worst pain imaginable. The distance from the left anchor point to the patient's mark will be measured and recorded.
pain score measured on VAS at time of tenaculum placemenet | collected at time of procedure.
  Level of pain at this step in the procedure will be recorded by patient on 100mm line where the left anchor point represents the absence of pain and the right anchor point represents the worst pain imaginable. The distance from the left anchor point to the patient's mark will be measured and recorded.
pain score measured on VAS at time of cervical dilation | collected at time of procedure.
  Level of pain at this step in the procedure will be recorded by patient on 100mm line where the left anchor point represents the absence of pain and the right anchor point represents the worst pain imaginable. The distance from the left anchor point to the patient's mark will be measured and recorded.
overall pain scores will be measured on VAS at the conclusion of the procedure | collected at conclusion of procedure.
  Level of pain at this step in the procedure will be recorded by patient on 100mm line where the left anchor point represents the absence of pain and the right anchor point represents the worst pain imaginable. The distance from the left anchor point to the patient's mark will be measured and recorded at the conclusion of the procedure.
overall satisfaction with pain management will be measured on a 5 point Likert scale | collected at conclusion of procedure
  Likert scale assessing satisfaction will be based on scale from 0 to 4 where 0 equals very unsatisfied and 4 equals very satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, Principal Investigator — PPNYC
Locations (1):
- Planned Parenthood- Boro Hall, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided